CLINICAL TRIAL: NCT04224324
Title: The Effect of Pediatric Patient Temperament on Postoperative Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Stephen Kelleher, Anesthesiologist, Boston Children's Hospital
Other Study IDs: IRB-P00033445
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Emergence Delirium; Temperament
MeSH Terms: conditions — Emergence Delirium | interventions — Tonsillectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T & A patients: pediatric patients undergoing tonsillectomy and adenoidectomy
  Interventions: Procedure: Tonsillectomy and Adeniodectomy

INTERVENTIONS:
Procedure: Tonsillectomy and Adeniodectomy — pediatric patients undergoing tonsillectomy and adenoidectomy

SUMMARY:
The goal of this study is to determine if preoperative temperament is associated with postoperative pain, emergence agitation, emotional and behavioral changes, and overall parent satisfaction. This is a prospective observational study to assess preoperative temperament in pediatric patients undergoing tonsillectomy and adenoidectomy, gather demographic data, intraoperative data regarding surgical and anesthetic technique, and collect immediate postoperative data to assess pain, emergence agitation (EA), parental satisfaction as well as remote postoperative data to assess emotional and behavior changes. These data will be used to determine if patients with a specific temperament profile are more likely to experience increased pain, emergence agitation, emotional changes, and behavioral disturbances postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* undergoing Tonsil and/or Adenoid Removal at Boston Children's Hospital

Exclusion Criteria:

* history of prematurity
* major chronic medical conditions
* neurological impairment or developmental delay
* parents/guardians who do not speak English or are unable to understand the questionnaires

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients undergoing tonsillectomy and adenoidectomy at Boston Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 344 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Temperament | preoperative period
  Patient temperament based on the Children's Behavior Questionnaire. This is a 36 question temperament inventory completed by the caregiver. Items are scored on a scale from 1 to 7, where 1 is "extremely untrue" and 7 is "extremely true". Total scores are linked to temperament constructs of Surgency, Negative Affectivity, and Effortful Control.
Pain score | immediately post operative period
  Pain behavior to be recorded using numerical rating scale (NRS), FLACC scale or Wong Baker Faces scale as appropriate for age and developmental status. All of these scales are scored from 1-10 where higher scores indicate more pain.
emergence agitation | immediately post operative period
  Measured using the Pediatric Emergence Delirium Scale (PAED). Scored on a scale from 0-4 where total scores of 10 or greater at any time during Post Anesthesia Care Unit (PACU) stay are classified as experiencing agitation.
post hospital behavior changes | up to 4 weeks after surgery
  Measured using the Post Hospitalization Behavior Questionnaire. Questions are answered on a scale of 1-5, where 1 is less than before and 5 is more than before. Adverse behavioral outcomes to be defined as those patients who experienced behavioral changes at one or more standard deviations above the sample mean.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States